CLINICAL TRIAL: NCT04727424
Title: A Multicenter, Prospective, Adaptive, Double-blind, Randomized, Placebo-controlled Study to Evaluate the Effect of Fluvoxamine Plus Budesonide, Fluoxetine Plus Budesonide and Spirulin Platensis, in High Risk Patients With Mild COVID-19
Brief Title: Repurposed Approved and Under Development Therapies for Patients With Early-Onset COVID-19 and Mild Symptoms
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cardresearch (Other)
Collaborators: Cytel Inc. (Industry); McMaster University (Other); Fastgrants (Unknown); Eiger BioPharmaceuticals (Industry); RainWater Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TOGETHER_2
Record Dates: First submitted 2021-01-25; First posted 2021-01-27 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Covid19; SARS-Associated Coronavirus
Keywords: COVID-19; Randomized study; Fluvoxamine; Budesonide; Fluoxetine; Spirulin Platensis
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — Fluvoxamine; Fluoxetine

STUDY DESIGN:
Intervention Model Description: TOGETHER trial is a Multiplatform, adaptive trial started on 20 Jan 2021. This description is in allignment as per amendment seven with Brazilian National Ethics Committee final decision letter (letter# 5416996) issued on May 18, 2022.
  Patients with mild disease will be screened at primary and secondary care public health services and randomly allocated to one of three treatment arms in a 1:1:1:1 ratio, as per described in detail in approved protocol version 8.0 dated 12 APR 2022.
  1. Fluvoxamine + Budesonide
  2. Fluoxetine + Budesonide
  3. Spirulin Platensis
  4. Placebo
  We will use a centralized random allocation schedule, generated by computer and stratified by site and age.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigational medical product will be packaged in similar bottles by a third party who will keep the allocation confidential until the end of the study. The bottles will be sealed and identified as "Research Product with no commercial value" and coded. They will be randomly allocated among the participants using a centralized randomization system The research subjects, medical assistance, administrative and health staff will not have access to the contents of the bottles. All arms will have a placebo counterpart with same dose schedule.
  All planned Data and Safety Monitoring Board (DSMB) interim analysis will be blinded. If needed a unblinded statistician will be provided if DSMB decides to stop any arm. At the end of the study, or early termination as per DMSB interim analysis plan, the arms will then be identified.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fluvoxamine Maleate + Budesonide Inhalation powder (Active Comparator): Fluvoxamine 100 mg oral tablets:
  One tablet after randomization (Day 0) followed by 100 mg BID for the following 09 days PLUS
  Budesonide Inhalation powder 400 mcg capsule:
  One 400 mcg capsule (inhalation) after randomization (Day 0) followed by one puff of 400 mcg BID for the following 09 days
  Interventions: Drug: Budesonide Powder; Drug: Placebo
- Spirulin Platensis (Active Comparator): Spirulin Platensis 500mg oral tablets Two tablets right after randomization (day 0) followed by 1.000mg (two tablets) BID for the following 10 days.
  Interventions: Dietary Supplement: Spirulin Platensis; Drug: Placebo
- Fluoxetine + Budesonide Inhalation powder (Active Comparator): Fluoxetine 20 mg oral tablets:
  Two tablets right after randomization (Day 0) followed by 40 mg MID for the following 06 days PLUS
  Budesonide Inhalation powder 400 mcg capsule:
  One 400 mcg capsule (inhalation) right after randomization (Day 0) followed by one puff of 400 mcg BID for the following 06 days
  Interventions: Drug: Fluoxetine 20 MG; Drug: Placebo
- Placebo (Placebo Comparator): Placebo oral tablets (10-day schedule):
  Matching tablets started after randomization using the dosing regimen of 01 tablet every 12 hs starting at Randomization Day (Day 0) until end of Day 09 (total of 10 day schedule)
  PLUS
  Placebo Inhalation Therapy:
  One dosing (inhalation puff) right after randomization (Day 0) followed by one puff BID for the following 09 days
  OR
  Paracetamol (07-day schedule - active comparator):
  Paracetamol 500 mg tablets started after randomization using the dosing regimen of 01 tablet BID starting at Rand. Day (Day 0) until end of Day 06 (total of 07 days schedule - ANTICOV Arm)
  OR
  Matching tablets started after randomization using the dosing regimen of 02 tablets every 12 hs starting at Randomization Day (Day 0) until end of Day 09 (total of 10 day schedule)
  Interventions: Dietary Supplement: Spirulin Platensis; Drug: Budesonide Powder; Drug: Fluoxetine 20 MG

INTERVENTIONS:
Dietary Supplement: Spirulin Platensis — Two tablets every 12 hours since randomization through day 09 following randomization
  Arms: Placebo; Spirulin Platensis
Drug: Budesonide Powder — One Fluvoxamine tablet every 12 hours since randomization through day 09. PLUS
  01 Budesonide powder (inhalation) every 12 hours since randomization through day 09.
  Other Names: Fluvoxamine Maleate 100 MG [Luvox]
  Arms: Fluvoxamine Maleate + Budesonide Inhalation powder; Placebo
Drug: Fluoxetine 20 MG — Two Fluoxetine tablets every day starting just after randomization through day 07.
  PLUS
  01 Budesonide powder (inhalation) every 12 hours since randomization through day 07.
  Other Names: Budesonide powder
  Arms: Fluoxetine + Budesonide Inhalation powder; Placebo
Drug: Placebo — Placebo oral tablets (10-day schedule):
  Matching tablets started after randomization using the dosing regimen of 01 tablet every 12 hs starting at Randomization Day (Day 0) until end of Day 09 (total of 10 day schedule)
  PLUS
  Placebo Inhalation Therapy:
  One dosing (inhalation puff) right after randomization (Day 0) followed by one puff BID for the following 09 days
  OR
  Paracetamol (07-day schedule - active comparator):
  Paracetamol 500 mg tablets started after randomization using the dosing regimen of 01 tablet BID starting at Rand. Day (Day 0) until end of Day 06 (total of 07 days schedule - ANTICOV Arm)
  OR
  Matching tablets started after randomization using the dosing regimen of 02 tablets every 12 hs starting at Randomization Day (Day 0) until end of Day 09 (total of 10 day schedule)
  Arms: Fluoxetine + Budesonide Inhalation powder; Fluvoxamine Maleate + Budesonide Inhalation powder; Spirulin Platensis

SUMMARY:
The COVID-19 pandemic has been characterized by high morbidity and mortality, especially in certain subgroups of patients. To date, no treatment has been shown to be effective in patients with early-onset disease and mild symptoms. Experimental studies have demonstrated a potential anti-inflammatory role of Fluvoxamine, Fluoxetine, Budesonide and Spirulin Platensis in SARS-CoV-2 infections and observational studies have suggested a reduced complications in patients with COVID-19 disease.

DETAILED DESCRIPTION:
In December 2019 a series of viral pneumonia cases were reported in the city of Wuhan, China and a new subtype of coronavirus has been identified as the causative agent of this condition. On February 11, 2000 the disease has been characterized as COVID-19 and on March 11 the World Health Organization (WHO) declared a state of worldwide pandemic. On January 25, 2021 there are 98,794,942 cases and 2,124,193 documented deaths (global case-fatality ratio of 2.15%).

To date, no early treatment has been identified as effective in combating this disease which has been identified as with high morbidity and mortality. Epidemiological data suggest that despite development of vaccines we will have hundreds od thousands of cases in the next two years.

Thus, we propose the prospective, double-blinded, randomized evaluation of potential therapies against SARS-CoV2 and some clinical evidence derived from observational studies on reducing complications if used early on the disease, before inflammatory cascade is fully activated.

Important considerations on TOGETHER Adaptive Trial:

1. The Pegylated Lambda interferon arm was ended on early February 2022.
2. The Proposal of a new arm: Spirulin platensis.
3. The Modification on primary endpoints that will be effective only for new arms added to the trial (Spirulin platensis).

ELIGIBILITY:
A - Inclusion Criteria (except fluoxetine + budesonide and paracetamol arms):

1. Patients over 18 years old with the ability to provide free and informed consent
2. Acute Flu-Like symptoms < 07 days.
3. Patients with at least ONE enhancement criteria:

   1. The. Age > 50 years old (does not need any of the other criteria)
   2. Diabetes mellitus requiring oral medication or insulin
   3. Systemic arterial hypertension requiring at least 01 oral medication for treatment
   4. Known cardiovascular diseases (heart failure, congenital heart disease, valvular disease, coronary artery disease, cardiomyopathies under treatment, clinically manifest heart diseases with clinical repercussions)
   5. Symptomatic and/or treated lung disease (emphysema, fibrosing diseases)
   6. Patients with symptomatic asthma requiring chronic use of agents to control symptoms.
   7. Obesity, defined as BMI > 30 kg/m2 in weight and height information provided by the patient;
   8. Transplant patients
   9. Patient with stage IV chronic kidney disease or on dialysis.
   10. Patient with temperature measured at screening > 38º C.
   11. Patients with at least one of the following symptoms: Cough, Dyspnea, Ventilator-dependent chest pain or myalgias with limitation of daily activities (Criterion limited to 25% of randomizations)
   12. Immunosuppressed patients/using corticosteroid therapy (equivalent to a maximum of 10 mg of prednisone per day) and/or immunosuppressive therapy)
   13. Patients with a history of cancer in the last 5 years or currently undergoing oncological treatment
4. Patient with positive rapid test for SARS-CoV2 antigen performed on occasion of the screening or patient with a positive SARS-CoV2 diagnostic test within 07 days of the onset of symptoms.
5. Willingness to use the proposed investigative treatment and follow the protocol-related procedures foreseen in the research.
6. Signing the Free and Informed Consent Form before any research procedures

B - Inclusion criteria for the Fluoxetine + Budesonide combination arm (07 days of treatment - partnership with the "ANTICOV Consortium"):

1. Patients over 18 years of age with the ability to provide free and informed consent.
2. Patients treated at a Basic Health Unit of the Unified Health System (SUS) or patients treated at emergency care units of the SUS or supplementary medicine with an acute clinical condition compatible with COVID 19.
3. Patients over 18 years of age and a history of at least ONE of the following criteria.

   1. Diabetes mellitus, heart disease, chronic kidney disease, chronic obstructive pulmonary disease, cerebrovascular diseases or patients considered to be underweight or overweight according to the investigator's judgment (BMI ≤ 16 or BMI > 25).

      OR
   2. Individuals aged ≥ 60 years without co-morbidities.

      4) COVID-19 confirmed by molecular or antigenic test for SARS-CoV-2 within up to 24 hours prior to screening and a maximum of 2 days after sample collection.

      5) Viral syndrome with or without pneumonia and arterial O2 saturation > 94%.

      6) Signing the Free and Informed Consent Form before any research procedures.

      7) Willingness to use the proposed investigational treatment and follow the procedures provided for in the research.

Exclusion Criteria:

1. Negative diagnostic test for SARS-CoV2 associated with acute flu-like symptoms (patients with a negative test taken early and becoming positive a few days later are eligible, as long as they are < 07 days from the onset of flu-like symptoms);
2. Patients with an acute respiratory condition compatible with COVID-19 treated in the primary care network and with a decision to be hospitalized;
3. Patients with acute respiratory symptoms due to other causes;
4. Dyspnea secondary to other acute and chronic respiratory causes or infections (e.g. decompensated COPD, Acute bronchitis, Pneumonia other than viral, Primary pulmonary arterial hypertension);
5. Patients requiring hospitalization due to COVID-19 or SpO2 ≤ 93%.
6. Exclusion criteria applicable to the 7-day treatment arms:

   1. Abnormal findings on physical examination: Respiratory rate ≥ 25 irm; blood pressure < 90/ 60 mmHg or > 160/ 100 mmHg; Weight < 45 kg; recent episodes of vomiting in the last 24 hours or diarrhea > 3 episodes in the last 24 hours or serum potassium below 3.5 mEq/L.
   2. Serious injury to any organ that requires resuscitation and continuous treatment.
   3. Use of chronic systemic corticosteroid therapy with prednisone equivalent doses of > 40 mg/day
   4. Ongoing immunosuppressive treatment
   5. History of known pulmonary arterial hypertension or pulmonary fibrosis
   6. Patients previously vaccinated with two doses for SARS-CoV-2, with the last dose administered less than 180 days after screening; Patients with a single dose of Janssen SARS-CoV-2 vaccine received (except Janssen vaccine) and unvaccinated patients can participate regardless of the period.
   7. Use of serotonin reuptake inhibitors (all)
   8. Patients vaccinated for SARS-CoV-2 (complete vaccination - 02 doses) within 06 months of the last dose before randomization or patients who received a "booster" dose at any time before randomization.
   9. For any new antiviral included in the study, prior treatment with the antiviral, presence of contraindication to its use or concomitant intake of medication prohibited for its use.
   10. Enrolled in other clinical trials with unregistered medicines or with a registered medicine that may interact with any of the study PIs or contraindicated as concomitant treatment in the last 3 months before screening.
7. Exclusion criteria applicable to the 10-day treatment arm:

   A. Chronic use of serotonin reuptake inhibitors other than sertraline B. Chronic use of corticosteroid therapy with prednisone equivalent doses of > 40 mg/day
8. Exclusion criteria applicable to the 14-day treatment arm: Patients with phenylketonuria;
9. Continued use of monoamine oxidation inhibitors (MAOIs): Phenelzine, Tranylcypromine, Selegiline, Isocarboxazid, moclobemide;
10. Patients with severe psychiatric disorders - schizophrenia, uncontrolled bipolar disorders, major depression with suicidal ideation.
11. Pregnant or breastfeeding patients;
12. History of severe ventricular cardiac arrhythmia (Ventricular Tachycardia, recovered ventricular fibrillation patients) or Long QT Syndrome;
13. Known history of decompensated heart failure (NYHA III or IV), recent myocardial infarction (event < 90 days from screening), unstable angina, recent coronary bypass surgery (procedure < 90 days from screening), recent stroke ( event < 90 days from screening), symptomatic carotid disease, or mitral or aortic stenosis of moderate to severe intensity;
14. Surgical procedure or hospitalization planned (for other indications) to occur during treatment or up to 5 days after the last dose of study medication;
15. Current daily and/or uncontrolled alcohol consumption, which in the investigator's view could compromise participation in the study;
16. History of seizures in the last month or uncontrolled seizures;
17. Clinical history of moderate to severe hepatic impairment or liver cirrhosis with Child-Pugh classification C;
18. Patients with known severe degenerative neurological diseases and/or serious mental illnesses as assessed by the investigator;
19. Inability of the patient or representative to give consent or adhere to the procedures proposed in the protocol;
20. Any clinical conditions, including psychiatric conditions, which in the investigator's view could be an impediment to the use of research medications;
21. Known hypersensitivity and/or intolerance to Spirulin Platensis, Budesonide, Fluvoxamine and Fluoxetine;
22. Use of medications which have a known interaction with Spirulin platensis, Budesonide, Fluvoxamine and Fluoxetine;
23. Inability to use the medications and formulations provided for in this research;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender will be assumed as patient self-reported
Enrollment: 7819 (Estimated)
Dates: Start 2021-01-19 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of fluvoxamine + budesonide, fluoxetine + budesonide, Spirulin platensis in emergency care visits due to the worsening of COVID-19; | 28 days
  Evaluation of emergency visits due to progression of COVID-19 symptoms and/or ocmplications
Rate of fluvoxamine + budesonide, fluoxetine + budesonide, Spirulin platensis in changing the need for Hospitalization due to COVID-19 progression and related complications, including lower respiratory tract infection (LRTI) | 28 days
  Hospitalization due to COVID-19 progression and related complications
Rate of fluvoxamine + budesonide, fluoxetine + budesonide, Spirulin platensis in changing SPO2 ≤ 93% after randomization | 28 days
  Reduction of SPO2 ≤ 93% after randomization

SECONDARY OUTCOMES:
Time to clinical changes (up to 28 days of randomization), defined as greater than 50% symptoms changing in reference to baseline symptoms. | Randomization through day 28
  time to > 50% clinical symptoms changes as reported on baseline visit (self reported)
Time to clinical failure, defined as time to need for hospitalization due to the clinical progression of COVID-19 or associated complications. | Randomization through day 28
  Time to hospitalization
Number of days with respiratory symptoms since randomization | Randomization through day 28
  Days with symptoms
Rate of all-cause hospitalizations | Randomization through day 28
  All cause hospitalizations
Rate of COVID-19 related hospitalizations | Randomization through day 28
  COVID-19 hospitalizations
Number of days on Mechanical Ventilator | Randomization through day 28
  Number of days on mechanical Ventilator
Number of Days on Intensive Care Unit | Randomization through day 28
  Number of days on Intensive Care Unit
Number of days on hospitalizations | Randomization through day 28
  Number of days on Hospitalization
Health and Functioning after COVID-19 disease | Day 14 and Day 28
  Self evaluation of health functioning post COVID using Promis Global Health Score. Short term scale is a 10 item patient-reported questionnaire using response options as a 5-point and one 11 point rating scale. Higher scores means better global health.
Numbers of days with respiratory symptoms on WURSS-21 scale after randomization | Randomization through day 28
  Numbers of days with respiratory symptoms on WURSS-21 scale after randomization
Time to symptom resolution | randomization through day 28
  Time to improvement > 50% of baseline symptomatology based on WURSS-21 Scale.
Adherence of Study drug | Randomization through day 10
  Percentage of adherence on Study drug

CONTACTS AND LOCATIONS:
Overall Officials: Gilmar Reis, MD,PhD., Study Chair — Cardresearch - Cardiologia Assistencial e de Pesquisa; Edward J Mills, FRCP, Study Director — McMaster University
Locations (12):
- Brazil (12):
  - CARDRESEARCH - Cardiologia Assistencial e de Pesquisa, Belo Horizonte, Minas Gerais
  - City of Betim, Betim, Minas Gerais
  - City of Brumadinho, Brumadinho, Minas Gerais
  - Hospital e Maternidade Santa Rita, Contagem, Minas Gerais
  - City of Governador Valadares, Governador Valadares, Minas Gerais
  - City of Ibirité, Ibirité, Minas Gerais
  - City of Igarapé, Igarapé, Minas Gerais
  - Centro Universitário FIPMOC, Montes Claros, Minas Gerais
  - City of Nova Lima, Nova Lima, Minas Gerais
  - Universidade Federal de Ouro Preto, Ouro Preto, Minas Gerais
  - City of Santa Luzia, Santa Luzia, Minas Gerais
  - City of Sete Lagoas, Sete Lagoas, Minas Gerais

IPD SHARING:
Plan to Share IPD: Yes
Patient tables and main data.
Supporting Information: SAP
Time Frame: As of protocol termination
Access Criteria: Upon request

REFERENCES:
- [Background] Rayner CR, Dron L, Park JJH, Decloedt EH, Cotton MF, Niranjan V, Smith PF, Dodds MG, Brown F, Reis G, Wesche D, Mills EJ. Accelerating Clinical Evaluation of Repurposed Combination Therapies for COVID-19. Am J Trop Med Hyg. 2020 Oct;103(4):1364-1366. doi: 10.4269/ajtmh.20-0995. PMID 32828137
- [Background] Park JJH, Mogg R, Smith GE, Nakimuli-Mpungu E, Jehan F, Rayner CR, Condo J, Decloedt EH, Nachega JB, Reis G, Mills EJ. How COVID-19 has fundamentally changed clinical research in global health. Lancet Glob Health. 2021 May;9(5):e711-e720. doi: 10.1016/S2214-109X(20)30542-8. PMID 33865476
- [Background] Forrest JI, Rawat A, Duailibe F, Guo CM, Sprague S, McKay P, Reis G, Mills EJ. Resilient Clinical Trial Infrastructure in Response to the COVID-19 Pandemic: Lessons Learned from the TOGETHER Randomized Platform Clinical Trial. Am J Trop Med Hyg. 2022 Jan 7;106(2):389-393. doi: 10.4269/ajtmh.21-1202. PMID 34996047
- [Background] Reis G, Mills E. Fluvoxamine for the treatment of COVID-19 - Author's reply. Lancet Glob Health. 2022 Mar;10(3):e333. doi: 10.1016/S2214-109X(21)00588-X. No abstract available. PMID 35180413
- [Background] Thorlund K, Sheldrick K, Mills E. Molnupiravir for Covid-19 in Nonhospitalized Patients. N Engl J Med. 2022 Mar 31;386(13):e32. doi: 10.1056/NEJMc2201612. Epub 2022 Mar 16. No abstract available. PMID 35294804
- [Background] Park JJH, Detry MA, Murthy S, Guyatt G, Mills EJ. How to Use and Interpret the Results of a Platform Trial: Users' Guide to the Medical Literature. JAMA. 2022 Jan 4;327(1):67-74. doi: 10.1001/jama.2021.22507. PMID 34982138
- [Background] Jhuti D, Rawat A, Guo CM, Wilson LA, Mills EJ, Forrest JI. Interferon Treatments for SARS-CoV-2: Challenges and Opportunities. Infect Dis Ther. 2022 Jun;11(3):953-972. doi: 10.1007/s40121-022-00633-9. Epub 2022 Apr 21. PMID 35445964
- [Background] Park JJH, Dron L, Mills EJ. Moving forward in clinical research with master protocols. Contemp Clin Trials. 2021 Jul;106:106438. doi: 10.1016/j.cct.2021.106438. Epub 2021 May 14. PMID 34000408
- [Background] Park JJH, Ford N, Xavier D, Ashorn P, Grais RF, Bhutta ZA, Goossens H, Thorlund K, Socias ME, Mills EJ. Randomised trials at the level of the individual. Lancet Glob Health. 2021 May;9(5):e691-e700. doi: 10.1016/S2214-109X(20)30540-4. PMID 33865474
- [Background] Lee Z, Rayner CR, Forrest JI, Nachega JB, Senchaudhuri E, Mills EJ. The Rise and Fall of Hydroxychloroquine for the Treatment and Prevention of COVID-19. Am J Trop Med Hyg. 2021 Jan;104(1):35-38. doi: 10.4269/ajtmh.20-1320. PMID 33236703
- [Background] Dron L, Dillman A, Zoratti MJ, Haggstrom J, Mills EJ, Park JJH. Clinical Trial Data Sharing for COVID-19-Related Research. J Med Internet Res. 2021 Mar 12;23(3):e26718. doi: 10.2196/26718. PMID 33684053
- [Background] Dillman A, Park JJH, Zoratti MJ, Zannat NE, Lee Z, Dron L, Hsu G, Smith G, Khakabimamaghani S, Harari O, Thorlund K, Mills EJ. Reporting and design of randomized controlled trials for COVID-19: A systematic review. Contemp Clin Trials. 2021 Feb;101:106239. doi: 10.1016/j.cct.2020.106239. Epub 2020 Dec 3. PMID 33279656
- [Result] Reis G, Dos Santos Moreira-Silva EA, Silva DCM, Thabane L, Milagres AC, Ferreira TS, Dos Santos CVQ, de Souza Campos VH, Nogueira AMR, de Almeida APFG, Callegari ED, de Figueiredo Neto AD, Savassi LCM, Simplicio MIC, Ribeiro LB, Oliveira R, Harari O, Forrest JI, Ruton H, Sprague S, McKay P, Glushchenko AV, Rayner CR, Lenze EJ, Reiersen AM, Guyatt GH, Mills EJ; TOGETHER investigators. Effect of early treatment with fluvoxamine on risk of emergency care and hospitalisation among patients with COVID-19: the TOGETHER randomised, platform clinical trial. Lancet Glob Health. 2022 Jan;10(1):e42-e51. doi: 10.1016/S2214-109X(21)00448-4. Epub 2021 Oct 28. PMID 34717820
- [Result] Reis G, Dos Santos Moreira Silva EA, Medeiros Silva DC, Thabane L, Cruz Milagres A, Ferreira TS, Quirino Dos Santos CV, de Figueiredo Neto AD, Diniz Callegari E, Monteiro Savassi LC, Campos Simplicio MI, Barra Ribeiro L, Oliveira R, Harari O, Bailey H, Forrest JI, Glushchenko A, Sprague S, McKay P, Rayner CR, Ruton H, Guyatt GH, Mills EJ. Effect of early treatment with metformin on risk of emergency care and hospitalization among patients with COVID-19: The TOGETHER randomized platform clinical trial. Lancet Reg Health Am. 2022 Feb;6:100142. doi: 10.1016/j.lana.2021.100142. Epub 2021 Dec 14. PMID 34927127
- [Result] Reis G, Silva EASM, Silva DCM, Thabane L, Milagres AC, Ferreira TS, Dos Santos CVQ, Campos VHS, Nogueira AMR, de Almeida APFG, Callegari ED, Neto ADF, Savassi LCM, Simplicio MIC, Ribeiro LB, Oliveira R, Harari O, Forrest JI, Ruton H, Sprague S, McKay P, Guo CM, Rowland-Yeo K, Guyatt GH, Boulware DR, Rayner CR, Mills EJ; TOGETHER Investigators. Effect of Early Treatment with Ivermectin among Patients with Covid-19. N Engl J Med. 2022 May 5;386(18):1721-1731. doi: 10.1056/NEJMoa2115869. Epub 2022 Mar 30. PMID 35353979
- [Result] Reis G, Moreira Silva EAS, Medeiros Silva DC, Thabane L, Campos VHS, Ferreira TS, Santos CVQ, Nogueira AMR, Almeida APFG, Savassi LCM, Figueiredo-Neto AD, Dias ACF, Freire Junior AM, Bitaraes C, Milagres AC, Callegari ED, Simplicio MIC, Ribeiro LB, Oliveira R, Harari O, Wilson LA, Forrest JI, Ruton H, Sprague S, McKay P, Guo CM, Limbrick-Oldfield EH, Kanters S, Guyatt GH, Rayner CR, Kandel C, Biondi MJ, Kozak R, Hansen B, Zahoor MA, Arora P, Hislop C, Choong I, Feld JJ, Mills EJ, Glenn JS; TOGETHER Investigators. Early Treatment with Pegylated Interferon Lambda for Covid-19. N Engl J Med. 2023 Feb 9;388(6):518-528. doi: 10.1056/NEJMoa2209760. PMID 36780676
- [Result] Reis G, Mills EJ, Glenn JS. Pegylated Interferon Lambda for Covid-19. Reply. N Engl J Med. 2023 Jun 1;388(22):2108. doi: 10.1056/NEJMc2303519. No abstract available. PMID 37256990
- [Result] Reis G, Mills EJ. Ivermectin Treatment for Covid-19. Reply. N Engl J Med. 2022 Dec 15;387(24):e66. doi: 10.1056/NEJMc2207995. No abstract available. PMID 36516104
- [Derived] Reis G, Augusto Dos Santos Moreira Silva E, Carla Medeiros Silva D, Thabane L, Santiago Ferreira T, Vitor Quirino Dos Santos C, Paula Figueiredo Guimaraes Almeida A, Cancado Monteiro Savassi L, Dias de Figueiredo Neto A, Lanna Franca Reis L, Helena de Souza Campos V, Bitaraes C, Diniz Callegari E, Izabel Campos Simplicio M, Barra Ribeiro L, Oliveira R, Harari O, Forrest JI, Lat PK, Dron L, Thorlund K, Mills EJ. Effect of spirulina on risk of hospitalization among patients with COVID-19: the TOGETHER randomized trial. Am J Clin Nutr. 2024 Sep;120(3):602-609. doi: 10.1016/j.ajcnut.2024.06.016. Epub 2024 Aug 15. PMID 39232602
- [Derived] Reis G, Dos Santos Moreira Silva EA, Medeiros Silva DC, Thabane L, de Souza Campos VH, Ferreira TS, Quirino Dos Santos CV, Ribeiro Nogueira AM, Figueiredo Guimaraes Almeida AP, Cancado Monteiro Savassi L, de Figueiredo Neto AD, Bitaraes C, Cruz Milagres A, Diniz Callegari E, Campos Simplicio MI, Barra Ribeiro L, Oliveira R, Harari O, Wilson LA, Forrest JI, Ruton H, Sprague S, McKay P, Guo CM, Guyatt GH, Rayner CR, Boulware DR, Ezer N, Lee TC, McDonald EG, Bafadhel M, Butler C, Rodrigues Silva J, Dybul M, Mills EJ; TOGETHER Investigators. Oral Fluvoxamine With Inhaled Budesonide for Treatment of Early-Onset COVID-19 : A Randomized Platform Trial. Ann Intern Med. 2023 May;176(5):667-675. doi: 10.7326/M22-3305. Epub 2023 Apr 18. PMID 37068273